CLINICAL TRIAL: NCT06220812
Title: Functional Outcomes of Low Level Laser Versus Pulsed Electromagnetic Therapy in Children With Supracondylar Humeral Fracture
Brief Title: Different Modalities Interventions Post Supracondylar Humeral Fracture in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ezzat Abd El Mageid, M.Sc. in Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHF-LLL-PEMF
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Supracondylar Humeral Fracture in Pediatric
Keywords: SCHF- low level laser- pulsed electromagnetic field.

STUDY DESIGN:
Intervention Model Description: low level laser and pulsed electromagnetic field will be applied separated to different study groups of children with supracondylar humeral fracture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group A (Experimental): 20 children will receive designed physical therapy program in addition to low level laser
  Interventions: Device: low level laser ,pulsed electromagnetic field .
- study group B (Experimental): 20 children will receive designed physical therapy program in addition to pulsed electromagnetic field .
  Interventions: Device: low level laser ,pulsed electromagnetic field .

INTERVENTIONS:
Device: low level laser ,pulsed electromagnetic field . — LLL ,ASA via Alessandro Volta, 9 .36057 Arcugnano- Italy. With 905-nm wavelength, and maximum power output of 500 mW, laser spot of approximately 1 cm2 .
  PEMF, ASA, Easy teraza serie (ETS), Italy 2011, its code F9020087 and 230 its voltage.

SUMMARY:
the aim of the study is comparing the effects of LLLT and PEMFT on range of motion of elbow and radioulnar joint ,pain ,muscles strength of upper limb and hand function in children with post-operative type II and III supracondylar humeral fracture.

DETAILED DESCRIPTION:
intervention study describe the effects of low level laser and pulsed electromagnetic field in children with supracondylar humeral fracture . All children will be randomly classified by envelope method into two study groups of equal number. study group A and study group B. Both groups will receive designed physical therapy program, 20 minutes, 3 times per week for six weeks in addition to study group A will receive LLLT, 5 minutes and study group B will receive the same physical therapy program, in addition to PEMF, 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 6 to 10 years of both genders.
2. All subjects have unilateral extension type II and III supracondylar humeral fracture requiring closed reduction and percutaneous pinning (CRPP).
3. The study will be start immediately after removal the splint.
4. Children clinically and medically stable.
5. Children able to follow verbal commands.
6. Children sample will represent those children who enrolled in schools and other not yet.

   -

Exclusion Criteria:

The patients will be excluded if they have one of the following criteria;

1. Previous soft tissue injury at the same affected side of fracture.
2. Presence of associated fractures on the ipsilateral or contralateral upper limb.
3. Active infection near the fracture site.
4. Children with congenital or acquired skeletal deformities in the upper limbs.
5. Children with neurological deficits such as convulsions, involuntary movements, receiving muscle relaxants.

   -

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
pain measurement | six weeks post intervention.
  Numerical pain rating scale will be used to assess elbow pain intensity pre and post treatment in both groups.
Range of motion measurement | six weeks post intervention
  The 2- in-1 Digital Angle Ruler goniometer will be used to assess elbow and radio-ulnar joint ROM (flexion-extension -supination and pronation) pre and post treatment in both groups

SECONDARY OUTCOMES:
Hand function | six weeks post intervention
  Jebsen-Taylor Hand Function Test (JHFT) will be used to assess hand function pre and post treatment in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: General hospital Beni-Seuif Beni-seuif, Study Chair — generalhosbns@gmail.com
Locations (1):
- General Beni-Seuif Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mulpuri K, Hosalkar H, Howard A. AAOS clinical practice guideline: the treatment of pediatric supracondylar humerus fractures. J Am Acad Orthop Surg. 2012 May;20(5):328-30. doi: 10.5435/JAAOS-20-05-328. No abstract available. PMID 22553105
- [Background] Vaquero-Picado A, Gonzalez-Moran G, Moraleda L. Management of supracondylar fractures of the humerus in children. EFORT Open Rev. 2018 Oct 1;3(10):526-540. doi: 10.1302/2058-5241.3.170049. eCollection 2018 Oct. PMID 30662761
- See also: Related Info — https://journals.lww.com/jaaos/fulltext/2012/05000/aaos_clinical_practice_guideline__the_treatment_of.9.aspx